CLINICAL TRIAL: NCT04499820
Title: Effet d'Une supplémentation Par OMEGA3 Dans la rétinopathie diabétique
Brief Title: Effect of OMEGA3 Supplementation in Diabetic Retinopathy
Acronym: OMEDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OMEDIA
Record Dates: First submitted 2020-07-03; First posted 2020-08-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUTROF Group (Experimental): vitamin and DHA supplementation
  Interventions: Dietary Supplement: Nutrof
- MERALUT Group (Placebo Comparator): vitamin A, natural flavonoids, lutein and zeaxanthin and no DHA
  Interventions: Dietary Supplement: Meralut

INTERVENTIONS:
Dietary Supplement: Nutrof — DHA docosahexaenoic acid Omega 3s may be of interest in cases of retinopathies.
  Arms: NUTROF Group
Dietary Supplement: Meralut — vitamin A, natural flavonoids, lutein and zeaxanthin
  Arms: MERALUT Group

SUMMARY:
The main objective of this study is to evaluate the efficacy at 6 months of omega 3 supplementation on macular capillary density measured in optical coherence tomography angiography in patients with minimal or moderate non proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a leading cause of vision loss worldwide and is a major public health problem.

In Western countries, the prevalence of DR is estimated to be 35% in diabetic patients, while diabetic macular edema (DME) affects 5% of them.

Currently, apart from the balance of diabetes and other cardiovascular risk factors, no specific treatment is given for the minimal and moderate non-proliferative forms.

* DHA concentration in the retina can be modified according to the patient's diet.
* Minimal diabetic retinopathy does not currently benefit from specific treatment outside of diabetic control.
* Omega 3 are already known for their beneficial effects on the retina, brain and cardiovascular system but their effectiveness has not been tested on diabetic retinopathy.
* It is therefore a question of evaluating whether an omega 3 supplementation, at a dosage of 1000mg per day, can treat a minimal or moderate stage of diabetic retinopathy.

A study by Salavila et al. has shown that the intake of LCω3PUFA, via a Mediterranean diet, improved the stage of DR in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* For women of childbearing age, an effective method of contraception is introduced and monitored throughout their participation in the study.
* Diabetic microangiopathy: minimal to moderate nonproliferative diabetic retinopathy according to the ETDRS (EarlyTreatment of DiabeticRetinopathyStudy) classification.
* AV > 6/10
* One eye included. If both are affected, the eye with the poorer perfusion should be included.
* Affiliated to a social security scheme

Exclusion Criteria:

* < 18 years old.
* Pregnant or breastfeeding woman
* Other retinal pathologies that may interfere with the results (Patients previously treated with anti-VEGF, aflibercept or intra-vitreal corticosteroids, history of glaucoma, vitrectomy, retinal laser, epiretinal membrane), choroidal neo-vascularization, uveitis, retinal vascular occlusion, significant macular edema, macular thickness > 280 µm, Eyes with spherical equivalent greater than 8 Diopters, OCTA images not interpretable with many artifacts.)
* Hypersensitivity to any of the components of Nutrof or Meralut
* Taking the antivitamin k
* Known deficit in G6PD-
* History of renal lithiasis
* Kidney failure
* Immunosuppression
* Chronic Ethylism
* History of hepatopathy
* Intracranial tumor, intracranial hypertension
* Refusal to participate
* Patient participating in an intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
density of the deep capillary plexus in optical coherence tomography angiography (OCTA) | six months
  Macular vascularization consists of three interconnected capillary plexuses: the superficial capillary plexus (SCp) located at the level of the optic fibres and the intermediate (ICP) and deep (DCP) capillary plexuses located respectively at the level of the inner and outer part of the inner nuclear layer.16 OCTA is a non-invasive imaging method of retinal vasculature that allows a qualitative but mainly quantitative analysis of the capillary plexuses. A last parameter that could not be evaluated precisely with the old fluorescein and OCT angiography techniques. OCTA is performed without injection of intravenous contrast agent and has no side effects. Several studies have shown that PCP is the plexus most affected by non-perfusion areas in diabetic retinopathy.

SECONDARY OUTCOMES:
capillary plexus density in OCTA | six months
  capillary plexus density
area (mm²) of the central avascular zone in OCTA | six months
  area (mm²
Visual acuity measurement ETDRS | six months
  Visual acuity
Stage of diabetic retinopathy: minimal, moderate or severe | six months
  Each stage of retinopathy may be associated with some degree of diabetic macular edema; macular edema is classified as minimal, moderate or severe, depending on its location relative to the centre of the macula. It is considered severe when it reaches the centre of the macula.
  Non-proliferative diabetic retinopathy (NPDR, no neo-vessels) Minimal non-proliferative DR (some microaneurysms or punctiform hemorrhages).
  * Moderate nonproliferative DR (by exclusion if neither minimal nor severe DRNP)
  * Severe nonproliferative DR (or preproliferative DR): "4, 2, 1" rule (retinal hemorrhages in 4 quadrants and/or venous dilatations in 2 quadrants and/or AMIR in 1 quadrant)
central retinal thickness (µm) in the 2 groups at 6 months | six months
  central retinal thickness
cholesterol level: Low-density lipoprotein, High-density lipoprotein and total cholesterol | six months
  cholesterol leve
triglycerid level | six months
  triglycerid level
glycated haemoglobin (percent) | six months
  In diabetes, the higher the blood glucose level, the more glucose attaches to hemoglobin and the higher the level of glycated hemoglobin. It therefore indicates whether the blood glucose level was, on average, higher or lower during the 2 months prior to the test. Glycated haemoglobin is measured every 2-4 months. A small amount of blood is drawn from a vein or from the fingertip (micro-method).
  Glycated haemoglobin (HbA1c) is a fundamental criterion for blood sugar control. It is essential for assessing the risk of complications.
  9% Very high 7% Recommended 5% Normal
Diet questionnaire | six months
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Creteil, Créteil, Creteil, France

IPD SHARING:
Plan to Share IPD: No